CLINICAL TRIAL: NCT05329805
Title: Effect of Job Crafting Intervention Program on Harmonious Work Passion and Career Commitment Among Nurses: A Randomized Clinical Trial
Brief Title: Effect of Job Crafting Intervention Program on Harmonious Work Passion and Career Commitment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Port Said University (Other)
Responsible Party: Principal Investigator, Heba Emad Elgazar, lecture of nursing administraion, Port Said University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 31
Record Dates: First submitted 2022-03-31; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Nurse's Role
Keywords: Job crafting; harmonious work passion; career commitment

STUDY DESIGN:
Intervention Model Description: open-label, two-arm Randomized Control Trail (RCT)
Masking Description: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): Job crafting intervention
  Interventions: Behavioral: job crafting intervention
- control group (No Intervention): Regarding the control group, the participants will receive a simple educational booklet with one-session

INTERVENTIONS:
Behavioral: job crafting intervention — the participated nurses will receive session about job crafting followed by activity related to job crafting
  Arms: interventional group

SUMMARY:
effect of job crafting intervention program on nurses' job crafting behaviors, harmonious work passion and career commitment.

DETAILED DESCRIPTION:
the study aims to evulate the effectiveness ofjob crafting intervention program on nurses' job crafting behaviors, harmonious work passion and career commitment.

Hypotheses:

H1: Nurses participating in the job crafting intervention will report, post intervention, high level of job crafting behaviors compared with those nurse nurses in control group H2: Nurses participating in the job crafting intervention will report, post intervention, high level of harmonious work passion compared with those nurse nurses in control group H3: Nurses participating in the job crafting intervention will report, post intervention, high level of career commitment compared with those nurse nurses in control group this is RCT study among nurses work in EL-Nasar hospital, port said, Egypt

ELIGIBILITY:
Inclusion Criteria:

* licensed nurses who worked in direct contact with patients in their services
* had at least six month of experience in the nursing profession,
* agreed to participate in the study

Exclusion Criteria:

* participating in any intervention program within the last 12 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
measuring the change of the job crafting behavior of nurses | 3 months
  measuring changes occure in job crafting behaviors after applied job crafting intervention program to nurses. the researcher will use A 13-item Job Crafting Scale (Petrou et al., 2012) including three dimensions: seeking resources (6 items), seeking challenges (3 items), and reducing demandaftins (4 items). the minimum score is 13 and maximize score is 65. Higher scores indicate higher nurses job crafting level.

SECONDARY OUTCOMES:
Harmonious work passion | 3 months
  measuring changes occure in harmonious work passion after applied job crafting intervention program to nurses. the research will use A 7-item instrument of harmonious work passion created by Vallerand et al. (2003). the minimum score is 7 and maximium score is 49. Higher scores indicate greater harmonious work passion of nurses
career commitment | 3 months
  measuring changes occure in career commitment after applied job crafting intervention program to nurses using eight-item scale (Blau, 1985). higher score indicated higher career commitment. minimum score is 8 and high score is 40. Higher scores indicate higher levels of nurses' career commitment

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication will be shared to open data repository.
Supporting Information: Study Protocol
Time Frame: the data will be available after publishing the trail (expected in 2023)
Access Criteria: Open access